CLINICAL TRIAL: NCT07052773
Title: Blinded Retrospective Study to Clinically Validate the Accuracy of the Lung Cancer Detection System (LCDS) AI-based Decision Support Tool for Lung Cancer Low-Dose CT
Brief Title: Clinical Evaluation of the Lung Cancer AI-based Decision Support Tool in Low-Dose Lung CT
Acronym: GenMedAILCSD1
Status: Completed | Type: Observational
Sponsor: Genesis Medical AI (Industry)
Responsible Party: Sponsor
Other Study IDs: 0077-23-ASMC; privately funded (Other: Genesis Medical AI)
Record Dates: First submitted 2025-06-22; First posted 2025-07-07 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer Screening
Keywords: Lung Cancer Screening; Artificial Intelligence; Low-Dose Computed Tomography; Pulmonary Nodule Detection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective LDCT Scan Cohort: This cohort consists of 100 de-identified low-dose CT (LDCT) chest scans collected from individuals aged 50-79 years, with a ≥20 pack-year smoking history. These scans, acquired between 2018 and 2023 during routine lung cancer screening, include cases both with and without radiologically confirmed pulmonary nodules. The scans will be retrospectively evaluated by the AI-based Lung Cancer Detection System (LCDS).
  Interventions: Device: Lung Cancer Detection System (LCDS)

INTERVENTIONS:
Device: Lung Cancer Detection System (LCDS) — An AI-based decision support software designed to detect solid pulmonary nodules on LDCT chest scans. In this study, the LCDS is applied retrospectively to 100 previously acquired LDCT scans, and its performance is compared to a ground truth established by double-read radiologist reports with arbitration.

SUMMARY:
The goal of this observational study is to clinically validate the accuracy of an AI-based decision support tool-the Lung Cancer Detection System (LCDS)-for detecting lung nodules in asymptomatic adults aged 50-79 with a history of heavy smoking who underwent low-dose chest CT (LDCT) scans.

The main questions it aims to answer are:

* Can the LCDS accurately detect the presence of solid pulmonary nodules on LDCT scans, as measured by sensitivity and specificity?
* How does the LCDS's performance compare to existing AI systems using the Area Under the Curve-Receiver Operating Characteristic (AUC/ROC) Curve?

Researchers will compare the AI-based interpretations to a ground truth established by consensus among radiologists' double-readings to see if the LCDS can accurately classify cases as 'lung nodule presence' or 'lung nodule absence'.

Participants will:

* Have their de-identified LDCT scans (collected between 2018 and 2023) reviewed retrospectively.
* Be evaluated through the LCDS tool, which will classify cases based on lung nodule presence.

Contribute to performance evaluation using sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and ROC analysis.

ELIGIBILITY:
Inclusion Criteria:

* Undergone an LDCT scan between 2018 and 2023, while a diagnosis record exists.
* Age is between 50-79 years old.
* History of smoking at least a 20 pack-year smoking history and currently smoke or have quit within the past 15 years.

Exclusion Criteria:

* History of lung cancer: Subjects with a previous diagnosis of lung cancer may be excluded to ensure that the study focuses on detecting new cases or evaluating the progression of the disease.
* Prior lung nodule detection: Individuals who have previously undergone LDCT scans with documented lung nodules that required medical intervention may be excluded to avoid potential confounding factors in the analysis.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population in this study reflects the typical clinical screening cohort targeted by current lung cancer early detection guidelines and is suitable for evaluating the diagnostic accuracy of an AI-based decision support tool under real-world conditions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity of LCDS for Detection of Solid Pulmonary Nodules | Through study completion, an average of 1 year
  Proportion of true positive cases correctly identified by the AI-based Lung Cancer Detection System (LCDS) out of all subjects with radiologist-confirmed pulmonary nodules (Ground Truth).
Specificity of LCDS for Detection of Solid Pulmonary Nodules | Through study completion, an average of 1 year
  Proportion of true negative cases correctly identified by the LCDS out of all subjects without pulmonary nodules, as defined by the radiologist consensus ground truth.

SECONDARY OUTCOMES:
Area Under the ROC Curve (AUC) for LCDS Performance | Through study completion, an average of 1 year
  The area under the receiver operating characteristic (ROC) curve comparing AI classifications with the radiologist-defined ground truth for nodule detection.
False Positive Rate per Case | Through study completion, an average of 1 year
  The average number of false positive nodule detections made by the Lung Cancer Detection System (LCDS) per LDCT scan. A false positive is defined as a nodule detected by the AI system that was not confirmed by the radiologist-established ground truth.

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Makori, MD, Principal Investigator — Assuta Medical Center; Shay Cohen, MBA, Study Director — Genesis Medical AI
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the following reasons:
  * Medical imaging data sensitivity: The study involves low-dose CT (LDCT) chest scans containing highly sensitive medical imaging data that, despite de-identification efforts, may retain identifying characteristics inherent to medical images
  * Institutional privacy policies: Assuta Medical Center's data governance policies and patient consent frameworks do not permit external data sharing beyond the original study scope
  * Re-identification risk: Advanced imaging analysis techniques could potentially re-identify patients from anatomical features visible in CT scans, even after standard de-identification procedures Israeli privacy legislation: Compliance with Israeli Privacy Protection Law and healthcare data regulations that restrict sharing of patient-derived medical data Ethics Committee limitations: The original ethics approval and informed consent did not include provisions for data sharing.